CLINICAL TRIAL: NCT05211635
Title: Plan D- a Randomized Controlled Trial of Vitamin D Supplementation in Psychotic Disorders Including the Use of Digital Measures
Brief Title: Plan D- Vitamin D Supplementation in Psychotic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mari Nerhus, Consultant in Psychiatry MD PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (REK)-86434
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: vitamin D; 25(OH)D; processing speed; digit symbol coding; negative symptoms
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Placebo- controlled randomized 1:1 comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Vitamin D3 capsule 50 µg
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo capsule with identical appearance to the experimental drug
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — One capsule daily for 84 days
  Other Names: Divisun 2000 IE
  Arms: Vitamin D
Other: Placebo — One capsule daily for 84 days
  Arms: Placebo

SUMMARY:
Background: Impairment in cognitive processing speed is a consistent finding in schizophrenia spectrum disorder. Vitamin D deficiency is found to be significantly associated with reduced processing speed. In this study, we will investigate the effect from vitamin D supplementation on processing speed.

Objective: The primary objective is to investigate whether vitamin D supplementation is superior to placebo in improving processing speed.

The secondary objectives are to investigate whether vitamin D supplementation is superior to placebo in improving negative symptoms, social and physical activity.

Study design: Randomized placebo-controlled double blind trial. Study population: Men and women, aged 18-65 years, diagnosed with a schizophrenia spectrum disorder, in treatment for their disorder at the Division for Mental Health at Akershus university hospital.

Intervention: Participants will be randomized 1:1 to either vitamin D3 (50µg capsules) or placebo daily for 12 weeks. The medical product or placebo will be given in addition to treatment as usual.

Study measures: Cognitive tests, symptom assessments and blood sampling for vitamin D analyses will be performed at baseline and after 12 weeks intervention. During the 12 week intervention period the participants will use a smart phone application (MinDag) for self-report and an actigraph (MotionWatch 8 actigraph from CamNtech) for registration of physical activity.

Endpoints: Primary outcome is change in cognitive performance on the symbol coding test from the Brief assessment of Cognition in Schizophrenia (BACS). Secondary outcomes are change in performance on the the Category Fluency Test from the MATRICS Consensus Cognitive battery, change in negative symptoms from the clinician rated Brief negative symptom scale (BNSS), and change in self-reported negative symptoms from the scale Self-assessment of negative Negative Symptoms (SNS). Secondary outcomes also include change in self-reported social activities and change in actigraph registered physical activity.

Expected benefits for consumers and caregivers: The results from the study will indicate whether vitamin D supplementation could represent a beneficial treatment strategy for impaired processing speed and related symptoms.

DETAILED DESCRIPTION:
Background:

Vitamin D deficiency is considered a risk factor for schizophrenia spectrum disorders. The influence from vitamin D may be specifically important in the developing fetal brain. However, vitamin D deficiency is also found to be associated with symptom severity in established schizophrenia spectrum disorder, indicating that vitamin D also plays an important role in the adult brain. Our research group has found a strong association between low vitamin D levels and higher symptom burden of depressive- and negative symptoms, and associations between vitamin D deficiency and cognitive impairments, reduced processing speed in particular. Our results are in line with results from other studies. Symptoms of vitamin D deficiency per se involves motor fatigue and muscle weakness, and vitamin D is found to be crucial for the connectivity in neuronal circuits responsible for both locomotor-, emotional- and reward dependent behavior. Despite the strong associations between vitamin D deficiency and core features of schizophrenia spectrum disorders, very few intervention studies have been performed in schizophrenia samples.

The cognitive impairment of reduced processing speed is evaluated by standardized cognitive tests. The task could be to match symbols and letters by writing on a sheet of paper, to draw a pattern or solve a puzzle. The ability to perform will thus be dependent on the actual physical speed, the interaction between brain activity and body movements, i.e. psychomotor function, and cognition. In this study we will therefore investigate vitamin D's effect om cognitive processing speed and the effects on other outcomes related to psychomotor function. We will use both well-known clinical methods as well as new digital measures to measure potential effects.

Sociodemographic and diagnostic assessments:

Age, sex, cultural background, education level, work-, and civil status will be mapped by a structured interview and by information obtained from patient records. The Structured Clinical Interview for DSM-5 Disorders, Clinician Version (SCID-5 CV) will be used for diagnostic purposes. Current medication will be registered by interview or obtained from patient records.

MinDag Smart phone application:

Participants will be asked to use the smart phone application MinDag (MyDay) during the 12 week trial period, and download the app to their own smartphone. MinDag was developed by a team of clinical researchers at Norment in collaboration with the Web-app group at the Oslo University Center for Information Technology (USIT). The final version is now implemented at the Norment center. The app consists of daily self-reports covering activities/functioning, and a biweekly module assessing negative symptoms.

Actigraph:

The participants will also be asked to wear a MotionWatch 8 actigraph from CamNtech, which will yield continuous measures of body acceleration. Actigraphs have proven to be important ambulatory tools to obtain objective measures of sleep and activity. However the main focus for the use of the actigraph is to measure body acceleration, i.e. physical activity. The MotionWatch 8 is CE-marked, waterproof and has a battery lives of approximately 3 months. Actigraphs have successfully been used in studies of schizophrenia spectrum disorders to investigate sleep patterns and physical activity.

Medical product and placebo:

Vitamin D3 supplements as oral capsules will be used for supplementation, with a dosage of 50 microgram (= 2000IE) daily. This dosage have not been associated with negative effects in former intervention studies and is considered sufficient to ensure significant increase in S-25(OH)D. Norwegian Scientific Committee for Food and Environment has proposed 100 microgram (= 4000IE) daily as upper tolerable intake limit for vitamin D substitution. To make sure the study participants do not risk intoxication we have chosen to dosage the vitamin D supplementation with half the dosage for non- tolerable dose.

Vitamin D is considered as a food supplement, not a medical drug. The research protocol has been submitted to the Norwegian Medicines Agency, who has concluded that the project is not categorized as a medical drug study.

Vitamin D measurements:

S-25(OH)D is perceived as a satisfactory indicator of the vitamin D level in the body and is the metabolite that will be measured and used in the analyses. Serum concentration of 25(OH)D reflects both vitamin D produced from the skin and that obtained from food and supplements. The half-life of S-25(OH)D is several weeks and S-25(OH)D is perceived as a satisfactory indicator of the vitamin D level in the body.

Statistics:

The main analyses will be performed in IBM SPSS Statistics for investigating group differences (T-test, ANOVA and regression models will be used for this purpose), and change form baseline to follow up (mixed models will be the preferred analytic model here). The biostatistical work group at the Norment center will be conferred for the statistical analyses, for analyzing data from the app and actigraph in particular. Possible confounders known from the literature will be controlled for, such as gender, age, cultural background and current medication.

Sample size calculation:

We assume that the primary outcome (results from digit symbol coding) is a continuous variable with a normal distribution. Two independent clinical groups will be compared. In a similar sample (participants with a psychotic disorder), the results showed mean value 53.06 and standard deviation 11.26 in digit symbol coding for participants with vitamin D level ≥25 nmol/L and mean 45.65 and standard deviation 9.58 in participants with vitamin D level < 25 nmol/L. This was a significant difference with t-test, t=3.59 (95% confidence interval 3.35-11.47), p<0.001 and estimated effect size Cohen's d= 11.42. With significant level set to give a statistical power of 0.80 and alpha of 0.05 and with the same anticipated group differences in mean and standard deviations in the treatment group versus the placebo group, sample size calculation indicate that a number of 76 participants (N= 38 in each group) will be sufficient. However, we expect around 15 % drop out rate and we therefore aim to include 90 participants (N= 45 in each group).

User involvement:

This project has had active user involvement since the planning of the project. There has been regular meetings over the last year between the PI and the user representatives. The formulation of the written consent and information material for participants are developed in collaboration with the user representatives. The current research protocol has been presented to the user representatives and they have provided relevant feedback. They support the project and find the project relevant for the target group, particularly as the project can highlight a treatment for better well-being, as well as contributing to increased knowledge in the field.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, schizophreniform disorder or psychotic disorder not otherwise specified
* ability to give informed consent
* S-25(OH)D< 75nmol/L

Exclusion Criteria:

* psychotic symptoms with organic etiology
* severe mental retardation (IQ<70)
* hyperparathyroidism
* hypercalcemia
* renal failure (s-creatinine levels above 90µmol/L in women and above 105µmol/L for men)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Processing speed | 12 weeks
  Performance on the symbol coding test from the Brief assessment of Cognition in Schizophrenia (BACS). In this test, the participant is given a printed sheet with a key, linking a number to a nonsense symbol. In the same sheet a row with randomly assigned numbers appears. The participant is then asked to fill out the right corresponding symbol to each number based on the given key, as many as possible within 90 seconds. Measure: number of correct numerals (range: 0-110).

SECONDARY OUTCOMES:
Fluency | 12 weeks
  The category fluency from the MATRICS Consensus Cognitive battery (MCCB)
Negative symptoms | 12 weeks
  Clinician rated negative symptoms will be evaluated by The Brief Negative Symptom scale (BNSS). The BNSS is a 13-item instrument designed for clinical trials and measures these 6 domains: Anhedonia (includes items Intensity of pleasure during activities, Frequency of pleasure during activities, Intensity of Expected pleasure from future activities), Asociality (includes Asociality behavior, asociality Internal experience), Avolition (includes avolition behavior, Avolition Internal experience), Blunted affect (incudes Facial expression, Vocal expression, Expressive gestures), Alogia (Includes quantity of speech, Spontaneous elaboration). All the items in the BNSS are rated on a 7-point (0-6) scale, with anchor points generally ranging from the symptom's being absent (0) to severe (6). The BNSS scale show excellent psychometric properties, and is sensitive to treatment effects within a 12 week period.
Self-reported negative symptoms | 12 weeks
  The Self-assessment of negative Negative Symptoms (SNS). The questionnaire included in the application MinDag downloaded on the participant's own smartphones. The SNS includes of a 20 item questionnaire allowing patients to evaluate themselves on the five dimensions of negative symptoms (social withdrawal, diminished emotional range, alogia, avolition and anhedonia). Each item is scored as either 2 (strongly agree), 1 (somewhat agree), or 0 (strongly disagree). Biweekly reported during the 12 week intervention period. The scale has shown excellent sensitivity and specificity.
Social activity | 12 weeks
  Self reported time spent at school and work, work training, rehabilitation and/or treatment, doing physical activities, hobbies/ leisure activities, and time spent with other people physically and on the phone, internet and/or social media. Reported daily in the smartphone application MinDag in the evening module
Physical activity | 12 weeks
  Passive registration of body acceleration by the MotionWatch 8 actigraph from CamNtech. Continuous registration during the 12 week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Mari Nerhus, PhD, Principal Investigator — Akershus University Hospital and University of Oslo, NORMENT
Locations (1):
- Akershus University Hospital, Division of Psychiatry, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No